CLINICAL TRIAL: NCT01576614
Title: A Prospective Randomized Study on the Role of Off-shift Robotic Telerounding on the Collaboration Between Physicians and Nurses in the Surgical Intensive Care Unit
Brief Title: The Role of Off-shift Robotic Telerounding Between Physicians and Nurses in the Surgical Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-071
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Off-shift Robotic Telerounding
Keywords: Comparing telephone VS RTP in SICU rounding practices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Nurse-Physician Rounding by Phone: The SICU's practice involves daily morning team rounding at the bedside. The team includes the critical care attending physician (AP), surgical resident physician, and critical care nurse. The AP is physically present in the SICU during these rounds and for the hours between approximately 7am and 7pm. During off-shift hours (7pm-7am), the AP is available by phone as the "on-call" attending physician. In addition to this on-call availability, the standard of practice in SICU for years has been that the on-call physician proactively places a telephone call to the SICU at least once every evening to perform "telephone rounds" with the resident physician aeach SICU patient.
  Interventions: Behavioral: Remote physician rounding
- Nurse-Physican rounding by R T P: Remote Telepresence Robotics (RTP) is a form of telemedicine that enables a fast and direct face-to-face response by a physician, located remotely, and may sometime utilize a mobile robot.
  RTP provides the physician the ability to teleconference with patients and other healthcare providers using two way audio visual technology. The sophistication of these devices varies and can range from simple video conferencing to remote robotic control devices with audio visual conferencing capabilities. The "robotic" capabilities refer to ability of the physician to remotely direct or drive the device from one location to another.
  The technology allows clinical experts to provide the right care at the right time and has become an accepted standard of care when used under appropriate circumstances.
  Interventions: Behavioral: Remote physician rounding

INTERVENTIONS:
Behavioral: Remote physician rounding — Use of Remote physician rounding using Remote Telepresence Robotics
  Other Names: RTP; Remote Telepresence Rounding; Telemedicne; Robotic rounds

SUMMARY:
Hypothesis: The use of a mobile robotic telepresence system for off-hours rounding in the surgical intensive care unit has an impact on nurse-physician collaboration.

Study question: Does the addition of mobile video communication provided by RTP affect nurse-physician collaboration during off shift rounding in the surgical intensive care unit when compared to the more common clinical practice of off-shift rounding using the telephone?

DETAILED DESCRIPTION:
This is a mixed-method study, involving both surveys and ethnographic fieldwork. The research team will utilize the Collaboration and Satisfaction About Care Decisions (CSACD) survey instrument at regular intervals to assess nurse-physician collaboration. The instrument is validated and reliable and has been extensively tested. Permission was obtained to use the instrument. The ethnographic investigation will run concurrently and be performed by a doctoral student from Massachusetts Institute of Technology (MIT). No part of the study will involve patient intervention. The study will be conducted in the surgical intensive care unit (SICU).

The survey-based portion of the study is a prospective, randomized, crossover-controlled trial; it will generate ordinal data regarding nurse-physician collaboration and satisfaction. The ethnographic portion of the study will involve observation and interviews. The MIT student will engage in unobtrusive observational shadowing of APs and nurses throughout the study, and will formally interview each observed AP and nurse twice during the entire length of the study: once at the onset of the study, and once as the study draws to conclusion. This observational shadowing will include visits to the SICU. All participants will be consented for the study. Consent for and implementation of these methods will be undertaken in a manner consistent with current best research practice; extensive measures will be taken to protect staff confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Full time registered nursing staff
* Resident physicians and critical care attending physicians

Exclusion Criteria:

* Non-registered nursing staff

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Full time Nursing and Physician Staff providing rounding services in the Surgical Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Collaboration and Satisfaction Survey About Care Decisions using CSACD Scores | One Year
  This is a mixed-method study, involving both surveys and ethnographic fieldwork. The research team will utilize the Collaboration and Satisfaction About Care Decisions (CSACD) survey instrument at regular intervals to assess nurse-physician collaboration. The instrument is validated and reliable and has been extensively tested. Permission was obtained to use the instrument

CONTACTS AND LOCATIONS:
Overall Officials: Timothy N. Liesching, MD, Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Clinic, Burlington, Massachusetts, United States

REFERENCES:
- See also: Telemedicine provider — http://www.intouchhealth.com